CLINICAL TRIAL: NCT07193095
Title: Brief MORE: A Mindfulness Intervention For Chronic Musculoskeletal Pain
Brief Title: This Project is a Three-arm RCT Evaluating Two, Single-session Behavioral Interventions for Adults With Chronic Musculoskeletal Pain (CMP) -- 1) Brief Mindfulness-Oriented Recovery Enhancement (B-MORE) vs. Empowered Relief (ER) -- Relative to the Traditional 8-week Version of MORE.
Acronym: Brief Relief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00006036
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic pain; Brief intervention; Remote
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Mindfulness Oriented Recovery Enhancement (B-MORE) (Experimental): B-MORE is a 2-hour, single session adaptation of the traditional MORE program.
  Interventions: Behavioral: Brief Mindfulness Oriented Recovery Enhancement
- Empowered Relief (ER) (Experimental): ER is an evidence-based 2-hour single session intervention for chronic pain
  Interventions: Behavioral: Empowered Relief
- Mindfulness Oriented Recovery Enhancement (MORE) (Experimental): MORE is an 8-week evidence-based treatment for chronic pain.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement

INTERVENTIONS:
Behavioral: Brief Mindfulness Oriented Recovery Enhancement — B-MORE is a 2-hour, single session adaptation of the traditional MORE program.
  Arms: Brief Mindfulness Oriented Recovery Enhancement (B-MORE)
Behavioral: Empowered Relief — ER is an evidence-based 2-hour single session intervention for chronic pain.
  Arms: Empowered Relief (ER)
Behavioral: Mindfulness Oriented Recovery Enhancement — MORE is an 8-week evidence-based treatment for chronic pain.
  Arms: Mindfulness Oriented Recovery Enhancement (MORE)

SUMMARY:
Researchers at Florida State University are investigating how the length of treatment influences outcomes for individuals with chronic musculoskeletal pain. The goal is to identify the most effective balance between treatment duration and pain relief. There are three treatment conditions in this study: two different brief pain management trainings and one standard-length training. Participants will be randomized to either of the brief trainings, attending a single, 2-hour, online training session, in which a trained facilitator will teach pain management techniques that are backed by research. If randomized to receive the standard-length training, participants will attend eight, 2-hour, online training session over eight weeks, in which a trained facilitator will also teach research-backed pain management techniques. Short surveys will be required at seven different time points: before starting treatment, immediately after the pain-management training, and then 2, 6, 12, 24, and 36 weeks after the training.

ELIGIBILITY:
Inclusion Criteria:

* (1) having a chronic musculoskeletal pain condition, (2) average pain of ≥ 3 in the previous week, (3) willingness to engage with study assessments and interventions, (4) understanding English instructions fluently, and (5) being 18 and above.

Exclusion Criteria:

* (1) unable to consent because of physical or mental incapacity, (2) have previous, formal mindfulness training (e.g., MBSR) or previously receiving Empowered Relief, (3) have pain from a current cancer diagnosis or cancer-related treatment, (4) unstable illness that may interfere with treatment, (5) had surgery within the previous three months, and (6) had pain relieving injections, such as cortisone or hyaluronate, within the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 6 months
  Recruitment feasibility will be assessed via total enrollment and randomization numbers within the first 6 months of the study. Study team projects that it will be feasible to recruit and randomize 30 adults with CMP within 6 months.
Treatment Adherence & Acceptability | From baseline to 9-month follow-up
  Adherence (percentage of total treatment time attended) will be better for the single-session interventions, but all three conditions will be rated as highly acceptable (as measured by the Theoretical Framework of Acceptability; TFA).

SECONDARY OUTCOMES:
PROMIS - Pain Intensity | From baseline to 9-month follow-up
  A 3-item questionnaire using a 5-point Likert-like scale (1- had no pain to 5- very severe). Questions include "In the past 7 days, How intense was your pain at its worst?"
PROMIS - Pain Interference | From baseline to 9-month follow-up
  An 8-item questionnaire using a 5-point Likert-like scale (1- not at all to 5- very much). Questions include "In the past 7 days, how much did pain interfere with work around the home?".

OTHER OUTCOMES:
PROMIS - Depression | From baseline to 9-month follow-up
  A 4-item questionnaire using a 5-point Likert-like scale (1- never to 5- very much). Statements include "In the past 7 days, I felt worthless."
PROMIS - Anxiety | From baseline to 9-month follow-up
  A 4-item questionnaire using a 5-point Likert-like scale (1- never to 5- almost always). Statements include "In the past 7 days, my worries overwhelmed me".
PROMIS - Sleep Disturbance | From baseline to 9-month follow-up
  A 6-item questionnaire using a 5-point Likert scale
World Health Organization - Quality of Life | From baseline to 9-month follow-up.
  A 2-question assessment to measure self-reported quality of life. Participants will be asked "How would you rate your quality of life?" with a 5-point Likert scale (with "1- very poor" to "5-very good"). Participants will also be asked "How satisfied are you with your health?" with a 5-point Likert like scale (with "1-very dissatisfied" to "5-very satisfied").
Brief Pain Catastrophizing Scale | From baseline to 9-month follow-up
  The Brief PCS is a validated, 6-item questionnaire on which participants rate their thoughts and feelings about pain on a 5-point Likert scale, ranging from 0 ("Not at all") to 4 ("All the time").
Five Facets of Mindfulness Questionnaire | From baseline to 9-month follow-up
  A validated, 15-item questionnaire assessing trait mindfulness. Questions include "I do jobs or tasks automatically without being aware of what I'm doing".
Savoring Beliefs Inventory | From baseline to 9-month follow-up
  A validated measure to assess positive savoring habits. Questions include "Before a good thing happens, I look forward to it in ways that give me pleasure in the present".
Mindful Reappraisal of Pain Sensations | From baseline to 9-months
  A validated, 9-item questionnaire assessing one's ability to mindfully reappraise arising pain sensations. Questions include "I "step back" from the pain and see it as something outside of me".
Acute Clinical Effects of Treatment Sessions | Immediately before and after each training session.
  Acute pain intensity, pain unpleasantness, anxiety, and desire for pain medication will all be measured via a 0-10 numeric rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Building B, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request from qualified individuals.